CLINICAL TRIAL: NCT01518348
Title: Clinical Evaluation of T.R.U.E. TEST Panel 3.2 in Children and Adolescents
Acronym: PREAII
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study has been updated with new protocol number
Sponsor: Allerderm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Mekos 107P3.2 401
Record Dates: First submitted 2011-03-16; First posted 2012-01-26 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Contact Dermatitis
Keywords: Patch Test; Contact Dermatitis; Allergy; Children; PREA
MeSH Terms: conditions — Dermatitis, Contact; Hypersensitivity | interventions — Patch Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patch Test (Experimental)
  Interventions: Biological: Patch Test

INTERVENTIONS:
Biological: Patch Test — Patch Tested with Gold sodium thiosulfate, 0.075 mg/cm2 in hydroxypropylcellulose · Hydrocortisone-17-butyrate, 0.020 mg/cm2 in polyvinylpyrrolidone· Methyldibromoglutaronitrile, 0.0053 mg/cm2 in polyvinylpyrrolidone·Bacitracin, 0.60 mg/cm2 in hydroxypropylcellulose· Parthenolide, 0.0030 mg/cm2 in polyvinylpyrrolidone· Disperse blue 106, 0.050 mg/cm2 in polyvinylpyrrolidone· Bronopol, 0.25 mg/cm2 in polyvinylpyrrolidone
  Other Names: T.R.U.E. TEST

SUMMARY:
To evaluate the diagnostic performance (primary) and safety (secondary) of seven T.R.U.E. Test Panel 3.2 allergens: Gold sodium thiosulfate, Hydrocortisone-17-butyrate, Bacitracin, Parthenolide, Methyldibromoglutaronitrile, Disperse blue 106, and Bronopol in pediatric subjects 6-18 years of age with suspected contact dermatitis based on symptoms and clinical history.

DETAILED DESCRIPTION:
The study population will include at least 100 consecutive subjects 6-17 years of age with suspected contact dermatitis based on symptoms and clinical history. Study subjects must be otherwise healthy and fulfill entry criteria.

Visit 1 (Day 0): Informed Consent, Inclusion/Exclusion Criteria Assessment, Medical and Medicine History, Pregnancy Test (for female subjects of child-bearing potential), Panel Placement.Visit 2 (Day 2): Panel Removal, Panel Adhesion and Irritation Assessment, AE and Concomitant Medication Review.Visit 3 (Day 3- approximately 72 hours after placement): Skin Reactions Assessed and Scored. Adverse Event and Concomitant Medication Review.Visit 4 (Day 4 approximately 96 hours after placement): Skin Reactions Assessed and Scored. Adverse Event and Concomitant Medication Review.Visit 5 (Day 7±1): Skin Reaction Assessed and Scored. AE and Concomitant Medication Review. Visit 6 (Day 21±2): Skin Reaction Assessed and Scored. AE and Concomitant Medication Review. Visit performed via phone call, unless investigator determines that subject should be seen in clinic.

Primary Endpoint: Frequency and characterization of positive reactions per allergen. Secondary Endpoint: Prevalence of late or persistent reactions, irritation, adhesion, subject-reported itching or burning, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and history potentially consistent with allergic contact dermatitis based on symptoms and clinical history (i.e., subjects are visiting the clinic/physician to diagnose, treat or resolve this condition).
* Children and adolescents 6 to 18 years of age, and in general good health.
* Adolescent females 15 years of age or older (or with menarche) must consent to a urine pregnancy test; urine test results must be negative for study inclusion.
* Informed consent must be signed and understood by subject. If under age, informed consent must be signed and understood by parent or legal guardian, consistent with all institutional, local and national regulations.

Exclusion Criteria:

* Topical corticosteroid treatment during the last 7 days on or near the test area.
* Systemic treatment with corticosteroids or other immunosuppressives during the last 7 days.
* Subjects currently receiving (or received during the previous 3 weeks) other investigational drugs, treatments or devices, or participating in another clinical study.
* Treatment with ultraviolet (UV) light (including tanning) during the previous 3 weeks.
* Acute dermatitis outbreak or dermatitis on or near the test area on the back.
* Subjects unable to comply with activity restrictions (e.g., protecting test panels from excess moisture due to showering or vigorous activity).
* Subjects unable or unwilling to comply with multiple return visits.
* Female subjects 15 years of age (or with onset of menarche) and older unable to consent to a urine pregnancy test, or those with a positive pregnancy test.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in Frequency and characterization of positive reactions per allergen. | 72 hours, 96 hours, 1 week, 21 Days

SECONDARY OUTCOMES:
Prevalence of late or persistent reactions, irritation, adhesion, subject-reported itching or burning, and adverse events. | 72 hours, 96 hours, 1 week, 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Cory Dunnick, MD, Principal Investigator — Anschutz Health and Wellness Center, University of Colorado, Aurora, Colorado; Joseph Fowler, MD, Principal Investigator — Dermatology Specialists, Louisville, KY
Locations (2):
- United States (2):
  - Anschutz Health and Wellness Center, University of Colorado, Aurora, Colorado
  - Dermatology Specialists, Louisville, Kentucky